CLINICAL TRIAL: NCT03286816
Title: The Effect of Intravenous Lactate Administration on Brain Lactate Concentrations and pH During Euglycemia and Hypoglycemia in Patients With Type 1 Diabetes With and Without Impaired Awareness of Hypoglycemia
Brief Title: The Effect of Intravenous Lactate on Brain Lactate Concentrations During Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Diabetes Research Foundation (Other); European Foundation for the Study of Diabetes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Lac_iv
Record Dates: First submitted 2016-11-23; First posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2016-11

CONDITIONS: Type 1 Diabetes Mellitus With Hypoglycemia
Keywords: type 1 diabetes mellitus; impaired awareness of hypoglycemia; lactate; MR spectroscopy
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sodium Lactate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactate infusion (Experimental): Subjects will receive an intravenous lactate infusion to elevate plasma lactate levels
  Interventions: Drug: Sodium Lactate
- NaCl infusion (Placebo Comparator): As a control condition, subjects will receive intravenous NaCl infusion
  Interventions: Drug: SodiumChloride

INTERVENTIONS:
Drug: SodiumChloride
  Arms: NaCl infusion
Drug: Sodium Lactate
  Arms: Lactate infusion

SUMMARY:
Patients with type 1 diabetes (T1DM) who are unable to perceive symptoms of hypoglycemia, referred to as impaired awareness of hypoglycemia (IAH), are at very high risk of severe hypoglycemia. IAH affects approximately 25% of patients with T1DM. Brain lactate may be involved in the development of IAH. A recent study indicated increased brain lactate utilization during hypoglycemia in T1DM patients with IAH, which did not occur in patients with normal awareness of hypoglycemia (NAH). Conversely, administration of lactate to patients with NAH has been shown to attenuate counterregulatory hormone responses to and symptomatic awareness of hypoglycemia, thus causing a situation that resembles IAH. It has, however, not been demonstrated whether the excess of lactate is actually taken up or metabolized by the brain, and if so whether this occurs under euglycemic or hypoglycemic conditions or both.

This project consists of two related studies. The objective of part 1 is to investigate the effect of elevated plasma lactate levels that are sufficient to impair awareness of hypoglycemia on brain lactate concentrations during euglycemia and hypoglycemia in T1DM patients with NAH. The objective of part 2 is to compare the effect of exogenous lactate on brain lactate concentrations between T1DM patients with NAH and T1DM patients with IAH.

Furthermore, this study aims to determine the effect of acute hypoglycemia on the inflammatory function and composition of peripheral blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes duration ≥ 1 year
* Age: 18-50 years
* Body-Mass Index: 18-30 kg/m2
* HbA1c: 42-75 mmol/mol (6-9%)
* Outcome Clarke questionnaire: 0-1 or >=3
* Blood pressure: <160/90 mmHg

Exclusion Criteria:

* Inability to provide informed consent
* Use medication other than insulin, except for oral contraceptives or stable thyroxin supplementation therapy
* Presence of any other medical condition that might interfere with the study protocol, such as brain injuries, epilepsy, a major cardiovascular disease event, known liver disease, anxiety disorders or a history of panic attacks.
* Microvascular complications of T1DM: Proliferative retinopathy, Symptomatic diabetic neuropathy (including autonomic neuropathy), Nephropathy; clinical/overt albuminuria or an estimated glomerular filtration rate <60ml/min/1.73m2
* MR(I) contraindications (pregnancy, severe claustrophobia, metal parts in body)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
the effect of intravenous lactate administration, compared to placebo, on brain lactate concentrations during euglycemia and hypoglycemia in patients with T1DM and normal awareness of hypoglycemia | during stable euglycemia (40 min) and hypoglycemia (45 min)
the effect of exogenous lactate on brain lactate concentrations during euglycemia and hypoglycemia between T1DM patients with normal awareness of hypoglycemia and T1DM patients with impaired awareness of hypoglycemia | during stable euglycemia (40 min) and hypoglycemia (45 min)

SECONDARY OUTCOMES:
The changes in counterregulatory hormone and to hypoglycemia in response to lactate infusion, compared to placebo, in patients with normal awareness of hypoglycemia | during stable euglycemia (40 min) and hypoglycemia (45 min)
The changes in and symptoms to hypoglycemia in response to lactate infusion, compared to placebo, in patients with normal awareness of hypoglycemia | during stable euglycemia (40 min) and hypoglycemia (45 min)
The changes in brain pH in response to intravenous lactate administration, compared to placebo | during stable euglycemia (40 min) and hypoglycemia (45 min)
Changes in immune cell composition capacity in response to hypoglycemia compared to euglycemia and in response to lactate infusion compared to placebo | during stable euglycemia (40 min) and hypoglycemia (45 min)
Changes in immune cell cytokine production capacity in response to hypoglycemia compared to euglycemia and in response to lactate infusion compared to placebo | during stable euglycemia (40 min) and hypoglycemia (45 min)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud umc, Nijmegen, Netherlands

REFERENCES:
- [Background] De Feyter HM, Mason GF, Shulman GI, Rothman DL, Petersen KF. Increased brain lactate concentrations without increased lactate oxidation during hypoglycemia in type 1 diabetic individuals. Diabetes. 2013 Sep;62(9):3075-80. doi: 10.2337/db13-0313. Epub 2013 May 28. PMID 23715622
- [Background] Veneman T, Mitrakou A, Mokan M, Cryer P, Gerich J. Effect of hyperketonemia and hyperlacticacidemia on symptoms, cognitive dysfunction, and counterregulatory hormone responses during hypoglycemia in normal humans. Diabetes. 1994 Nov;43(11):1311-7. doi: 10.2337/diab.43.11.1311. PMID 7926305
- [Background] Maran A, Crepaldi C, Trupiani S, Lucca T, Jori E, Macdonald IA, Tiengo A, Avogaro A, Del Prato S. Brain function rescue effect of lactate following hypoglycaemia is not an adaptation process in both normal and type I diabetic subjects. Diabetologia. 2000 Jun;43(6):733-41. doi: 10.1007/s001250051371. PMID 10907119
- [Background] Wiegers EC, Rooijackers HM, Tack CJ, Heerschap A, de Galan BE, van der Graaf M. Brain Lactate Concentration Falls in Response to Hypoglycemia in Patients With Type 1 Diabetes and Impaired Awareness of Hypoglycemia. Diabetes. 2016 Jun;65(6):1601-5. doi: 10.2337/db16-0068. Epub 2016 Mar 18. PMID 26993070
- [Derived] Wiegers EC, Rooijackers HM, van Asten JJA, Tack CJ, Heerschap A, de Galan BE, van der Graaf M. Elevated brain glutamate levels in type 1 diabetes: correlations with glycaemic control and age of disease onset but not with hypoglycaemia awareness status. Diabetologia. 2019 Jun;62(6):1065-1073. doi: 10.1007/s00125-019-4862-9. Epub 2019 Apr 19. PMID 31001674